CLINICAL TRIAL: NCT03648034
Title: Effects of Preoperative Scalp Nerve Block on Postoperative Recovery Quality in Patients Undergoing Excision of Intracranial Meningioma
Brief Title: Effects of Scalp Nerve Block With Ropivacaine on Postoperative Recovery Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jie Tian, Principal Investigator, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SNB20180813
Record Dates: First submitted 2018-08-13; First posted 2018-08-27 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ropivacaine (Experimental): After anesthesia induction but before skull-pin insertion, patients in this group will receive scalp nerve blocks with 0.5% ropivacaine
  Interventions: Procedure: ropivacaine
- saline (Placebo Comparator): After anesthesia induction but before skull-pin insertion, patients in this group will receive scalp nerve blocks with 0.9% saline
  Interventions: Procedure: saline

INTERVENTIONS:
Procedure: ropivacaine — To perform scalp nerve blocks with ropivacaine
  Arms: ropivacaine
Procedure: saline — To perform scalp nerve blocks with saline
  Arms: saline

SUMMARY:
Patients undergoing elective meningeoma resection surgery will be randomly assigned to one of the following two groups. After anesthesia induction but before skull-pin insertion, one group will receive scalp nerve blocks with 0.5% ropivacaine, whereas the other group will receive scalp nerve blocks with 0.9% saline. The patients' postoperative recovery quality, which is evaluated by KPS score, peri-operative inflammatory responses, and post-operative pain degree will be evaluated and compared between the two groups.

DETAILED DESCRIPTION:
Patients undergoing elective meningeoma resection surgery will be randomly assigned to one of the following two groups. After anesthesia induction but before skull-pin insertion, one group will receive scalp nerve blocks with 0.5% ropivacaine, whereas the other group will receive scalp nerve blocks with 0.9% saline. The patients' KPS scores at 3d after surgery and at discharge, serum levels of TNF-α、IL-6，IL-1β at 24h after surgery, satisfaction score after recovery, and VAS scores at 1, 2, 3 days post-surgery will be evaluated and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. BMI 18-28 kg/m2;
3. ASA Physical Status 1-2;
4. Clinical diagnosis of primary Meningeoma and will have elective Meningeoma Resection Surgery;
5. With an estimated surgery time of less than 4h;
6. The incision will be conducted at the frontal, top or the temperal skull.

Exclusion Criteria:

1. A history of previous brain surgery;
2. Severe systemic disease (heart, lung, kidney, or immune system);
3. Nerval or mental disorders;
4. A history of addiction to opioids;
5. Allergic to ropivacaine;
6. Infection at block site or severe systemic infection;
7. Refuse to attend the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
KPS score | 7 days post-surgery
  Karnofsky performance score (KPS) allows patients to be classified as to their functional impairment. The total scale range is 0-100. The lower the KPS score, the worse the survival for most serious illnesses.

SECONDARY OUTCOMES:
KPS score | 3 days post-surgery
  Karnofsky performance score (KPS) allows patients to be classified as to their functional impairment. The total scale range is 0-100. The lower the KPS score, the worse the survival for most serious illnesses.
serum TNF-α levels | at 1h and 24h post-surgery
  an inflammatory mediator that reflects systemic inflammation
serum IL-6 levels | at 1h and 24h post-surgery
  an inflammatory mediator that reflects systemic inflammation
serum IL-1β levels | at 1h and 24h post-surgery
  an inflammatory mediator that reflects systemic inflammation
Iowa Satisfaction with Anesthesia Scale (ISAS) | 1 hour after the surgery is finished
  Iowa Satisfaction with Anesthesia Scale (ISAS) comprises of 11 items to measure patient satisfaction after surgery. The total scale range is -33-+33. The higher the ISAS score, the better the satisfaction level.
white blood cell | at 24 h after surgery
  serum white blood cell count
serum levels of CRP | at 24 h after surgery
  inflammatory responses
VAS score | at 1, 2 and 3 days post-surgery
  The visual analogue scale or visual analog scale (VAS) measures the average intensity of pain in the past on a 0-to-10 scale, where 0 = No pain and 10 = Pain as intense as you can imagine.
pain-relief medications | at 1, 2 and 3 days post-surgery
  amounts of pain-relief medications
Hospitalization Days | up to 30 days
  length of hospitalization
out of pocket expenditure for hospitalisation | hospital discharge/up to 30 days
  This reflects how much money the patient spends during hospitalisation
complications | within 30 days after surgery
  incidence of intracranial infection

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital affliated to Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided